CLINICAL TRIAL: NCT04827940
Title: The Effect of Progressive Relaxation Exercise With Music Therapy on Sleep Quality and Pain Intensity of Patients Hospitalized in Surgical Services
Brief Title: The Effect of Progressive Relaxation Exercise With Music Therapy on Sleep Quality and Pain Intensity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Pınar Duru, assistant professor, Eskisehir Osmangazi University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 25403353-050.99-E.27718
Record Dates: First submitted 2021-03-28; First posted 2021-04-01 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Postoperative Pain; Postoperative Sleep Quality
Keywords: Pain; Postoperative; Sleep; progressive relaxation exercise; music
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Intervention Model Description: This single-blind, pre-test-post-test with control group design quasi-experimental study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention arm (Experimental): Data from the study was collected during the implementation of the "Nursing Surgical Diseases" class. Students who completed the 4-hour training program on sleep, relaxation exercises and survey practice have been pollsters of the study.
  Relaxing music for sleep, prepared by the Turkish Psychological Association, is uploaded to patients' mobile phones. Patients were asked to perform relaxation exercises for a week at bedtime, lasting an average of 30 minutes, and with music every day, taking advantage of nurse observation at the clinic with the patient's declaration in check. Students who took part in the practice served as reminders of patients' compliance with the exercises.
  Interventions: Other: Progressive relaxation exercise with music
- Control arm (Other): Those who did not do progressive muscle relaxation exercises or did not practice regularly for a week constituted the control group.
  Interventions: Other: Progressive relaxation exercise with music

INTERVENTIONS:
Other: Progressive relaxation exercise with music — The progressive relaxation technique includes exercises for the muscles in the body to consciously contract and relax together with deep breathing exercises while sitting comfortably or lying down accompanied by music.
  Relaxing relaxation music for sleep, prepared by the Turkish Psychologists Association, has been installed on the mobile phones of the patients.
  The patients did the relaxation exercises for an average of 30 minutes before going to bed for a week and every day with music.Relaxing relaxation music for sleep, prepared by the Turkish Psychologists Association, has been installed on the mobile phones of the patients.
  The patients were taught to do the relaxation exercises for an average of 30 minutes before going to bed for a week and every day with music.

SUMMARY:
This study was conducted to determine the effect of progressive relaxation exercises with music therapy on sleep quality and pain severity of patients hospitalized in the surgical departments of a university hospital.This single-blind, pre-test-post-test with control group design quasi-experimental study was carried out between March-July 2019. 31 patients who were hospitalized in surgical departments for at least one week and regularly performed relaxation exercises consisted of experimental group, and 31 patients who were hospitalized for at least one week but did not do relaxation exercises consisted of control group. The study data were collected by using "Descriptive Characteristics Form", pain severity of patients was measured using "Visual Analogue Scale", and sleep quality of patients was measured using "Visual Analogue Sleep Scale". The patients were asked to perform the exercises with music an average of 30 min before sleeping every day for a week. The observation of the nurse working in department and the patient's statement were used for control. The ethical permission and the approval of hospital management were obtained for the study. In the statistical analysis of the data, independent sample t test, one-way anova and paired sample t test were used. Statistical significance level was taken as p<.05.

DETAILED DESCRIPTION:
Inclusion criteria in the study:

* Agree to participate in research
* Staying in surgical wards for at least one week between the dates of the study
* Being 18 years or older
* Not regularly practicing relaxation exercises before

Exclusion criteria from the study:

* Refusing to participate in research
* Being discharged before one week after admission to surgical services within the range of the study date
* Those who are hospitalized for more than a week due to the possibility of serious illness diagnoses that prevent patients from performing relaxation exercises
* Being 18 years or younger
* Communication problem
* Regularly practicing previous relaxation exercises

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in research
* Lying in surgical wards for at least a week in the range of the date of the study
* Being 18 or older
* Don't practice relaxation exercises regularly before

Exclusion Criteria:

* Not agreeing to participate in research
* Discharge before a week after admission to surgical wards within the range of the date of the study
* Those with more than a week's sleep due to the likelihood that patients may have received serious disease diagnoses that would put them off doing relaxation exercises
* Being 18 and under
* Don't be a communication problem
* Practice relaxation exercises regularly before

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
postoperative pain | In two groups, pain intensity pre-test and post-test values were measured with Visual Analog Scale. Pre-tests were evaluated in the first hour of their arrival in the service. Post-tests were measured at 09.00 in the morning on the 7th postoperative .
  Incision site pain experienced after surgery
postoperative sleep quality | In two groups, sleep quality pre-test and post-test values were measured with Visual Analog Sleep Scale. Pre-tests were applied before the surgery. Post-tests were measured at 09.00 in the morning on the 7th postoperative
  Quality of sleep in hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Örsal, Dr., Study Chair — ESOGUOU; Nedime Köşgeroğlu, Dr., Study Chair — İstanbul Rumeli University
Locations (1):
- Eskişehir Osmangazi University Practice and Research Hospital, Eskişehir, Odunpazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No